CLINICAL TRIAL: NCT05771779
Title: A Co-administration Study of Oral Cholera Vaccine (OCV), Typhoid Conjugate Vaccine (TCV), Measles and Rubella (MR) Vaccines in Bangladesh
Brief Title: Co-administration Study of OCV, TCV and MR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-23003
Record Dates: First submitted 2023-02-15; First posted 2023-03-16 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-08

CONDITIONS: Typhoid; Cholera; Measles; Rubella
Keywords: Co-administration; Immunogenicity; Safety; Typhoid fever; Cholera; Measles and Rubella; Conjugate vaccine
MeSH Terms: conditions — Typhoid Fever; Cholera; Measles; Rubella | interventions — Cholera Vaccines

STUDY DESIGN:
Intervention Model Description: An open-label, randomized controlled, non-inferiority study of co-administration of OCV, TCV and MR vaccines among children 12 to 59 months of age in Dhaka, Bangladesh will be conducted. Children who did not receive any of the aforementioned vaccines will be included in the study.
Masking Description: This is a open-label, randomized controlled, non-inferiority study. Study investigators along with study staff involved in safety evaluation and laboratory analysis will be blinded regarding the assigned treatment of the participant. The vaccine administration team will be un-blinded to the treatment assignment list. The vaccine administrator team members will not be involved in the evaluation of vaccine safety and laboratory analysis. The DSMB will be responsible for un-blinding the randomization number codes in the event of severe putative vaccine reactions. Otherwise, the codes will not be revealed until the end of the trial and until the computerized dataset has been frozen. If the intervention assignment is un-blinded, all study collaborators will be notified immediately. If deemed necessary, the DSMBs will recommend unblinding to the IRB and contact the study statistician responsible for providing information on the vaccine received by the individual in question.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm A: Oral Cholera Vaccine (OCV) only (Experimental): Based on randomization (n= 413) Potential participants will be vaccinated with OCV on Day 0 and Day 28. Two doses of MR vaccine will be given on day 56 and day 236. A blood sample (2-3 ml) will be collected for immunological assay on Day 0, Day 28, Day 56, Day 84 and Day 264 . All details will be recorded in the eCRF.
  Interventions: Biological: Oral Cholera Vaccine (OCV); Biological: Measles and Rubella (MR)
- Arm B: Typhoid Conjugate Vaccine (TCV) only (Experimental): Based on randomization (n= 314) Potential participants will be vaccinated with TCV on Day 0 and two doses of MR vaccine will be given on Day 56 and Day 236. A blood sample (2-3 ml) will be collected for immunological assay on Day 0, Day 28, Day 84 and Day 264 . All details will be recorded in the eCRF.
  Interventions: Biological: Typhoid Conjugate Vaccine (TCV); Biological: Measles and Rubella (MR)
- Arm C: Measles and Rubella (MR) only (Experimental): Based on randomization (n= 250) Potential participants will be vaccinated with MR on Day 0 and Day 180. A blood sample (2-3 ml) will be collected for immunological assay on Day 0, Day 28 and Day 208 . All details will be recorded in the eCRF.
  Interventions: Biological: Measles and Rubella (MR)
- Arm D: Co-administration of Measles and Rubella (MR) and Typhoid Conjugate Vaccine (TCV) (Experimental): Based on randomization (n= 314) Potential participants will be vaccinated with TCV on Day 0 and two doses of MR vaccine will be given on Day 0 and Day 180 . A blood sample (2-3 ml) will be collected for immunological assay on Day 0, Day 28 and Day 208 . All details will be recorded in the eCRF.
  Interventions: Biological: Typhoid Conjugate Vaccine (TCV); Biological: Measles and Rubella (MR)
- Arm E: Co-administration of Measles and Rubella (MR) and Oral Cholera Vaccine (OCV) (Experimental): Based on randomization (n= 413) Potential participants will be vaccinated with OCV on Day 0 and Day 28 . Two doses of MR vaccine will be given on Day 0 and Day 180 . A blood sample (2-3 ml) will be collected for immunological assay on Day 0, Day 28 , Day 56 and Day 208 . All details will be recorded in the eCRF.
  Interventions: Biological: Oral Cholera Vaccine (OCV); Biological: Measles and Rubella (MR)
- Arm F: Co-administration of Typhoid Conjugate Vaccine (TCV) and Oral Cholera Vaccine (OCV) (Experimental): Based on randomization (n= 413) Potential participants will be vaccinated with TCV on Day 0 . Two doses of OCV vaccine will be given on Day 0 and Day 28. Also two doses of MR vaccine will be given on Day 56 and Day 236. A blood sample (2-3 ml) will be collected for immunological assay on Day 0, Day 28 , Day 56 , Day 84 and Day 264 . All details will be recorded in the eCRF.
  Interventions: Biological: Oral Cholera Vaccine (OCV); Biological: Typhoid Conjugate Vaccine (TCV); Biological: Measles and Rubella (MR)

INTERVENTIONS:
Biological: Oral Cholera Vaccine (OCV) — Bivalent, Killed, Whole Cell Oral Cholera Vaccine
  Arms: Arm A: Oral Cholera Vaccine (OCV) only; Arm E: Co-administration of Measles and Rubella (MR) and Oral Cholera Vaccine (OCV); Arm F: Co-administration of Typhoid Conjugate Vaccine (TCV) and Oral Cholera Vaccine (OCV)
Biological: Typhoid Conjugate Vaccine (TCV) — Vi-polysaccharide conjugated to tetanus toxoid, Vi-TT
  Arms: Arm B: Typhoid Conjugate Vaccine (TCV) only; Arm D: Co-administration of Measles and Rubella (MR) and Typhoid Conjugate Vaccine (TCV); Arm F: Co-administration of Typhoid Conjugate Vaccine (TCV) and Oral Cholera Vaccine (OCV)
Biological: Measles and Rubella (MR) — Live attenuated vaccine

SUMMARY:
An open-label, randomized controlled, non-inferiority study of co-administration of OCV, TCV and MR vaccines among children 12 to 59 months of age in Dhaka, Bangladesh will be conducted. Children who did not receive any of the aforementioned vaccines will be included in the study.

This study will be conducted among 2117 children of 12-59 months of age residing in Mirpur area (wards 4, and 6-16) of Dhaka north and Kamrangirchar, Hazaribag and Rayerbazar areas (wards 14, 22, 56, 57, and 58) of Dhaka south to enroll the required number of participants. Only children who have not previously received the vaccines will be enrolled. The findings of this study are likely to have a significant impact on vaccine co-administration strategies for campaign and routine immunization programs. The participants will be randomly assigned to one of the six arms. The numbers are defined for each arm based on the sample size calculation. A list of children who did not receive MR, OCV and TCV will be prepared before enrollment by trained study staff (TSS). The TSSs will visit households in the defined study area and ask if the parents/guardians of children aged 12-59 months are willing to participate in the study. If they show willingness to participate, the TSSs will check their vaccination cards (if available) and prepare the list of potentially eligible children who have not received OCV, TCV and MR based on their vaccination card status and verbal statement (if vaccination card is not available). The investigators will enroll the participants after obtaining informed written consent and collect around 2-3 ml blood from each participant at different time points.

DETAILED DESCRIPTION:
The investigators will use an open-label, randomized controlled study design, to assess potential interference of antibody responses for different combinations of vaccines such as MR+TCV, MR+OCV and OCV+TCV. The study will be conducted among children aged 12-59 months in areas of urban Dhaka Bangladesh. Children will eligible for inclusion if they had not previously received OCV, TCV and MR.

Hypothesis:

Seroconversion following co-administration of OCV, TCV and MR at different combinations is non-inferior to seroconversion following administration of the vaccines alone.

Study activities:

Screening and eligibility assessment:

Study staff will invite participants to the field offices to be enrolled in the study. If agreed, written consent will be obtained from the parent/guardian at the field office. Clinical assessment will be done. After screening, the eligible participant will be enrolled for vaccination in different arms after matching with eligibility criteria. A study ID will be provided to each participant once informed written consent has been obtained.

Informed consent The parent/guardian must personally sign and date the latest approved version of the informed consent form before any trial specific procedures are performed. The parent/guardian will be provided with a copy of the signed consent form for their retention.

Enrollment Potential participants will attend the vaccination site. Upon arrival, inclusion/exclusion criteria will be assessed. Physical examination will be carried out prior to vaccination. The participant will then be vaccinated by oral cholera vaccine (OCV), Euvichol-Plus against V. cholerae; typhoid conjugate vaccine (TCV), Typbar-TCV for S. Typhi; MR vaccine for measles and rubella and a blood sample (2-3 ml) will be collected for immunological assay before vaccination. All details will be recorded in the eCRF. Based on the randomization of the six arms (mention below), the appropriate vaccine will be administered by a trained study staff (TSS).

Six study arms:

Arm A: OCV only Arm B: TCV only Arm C: MR only Arm D: Co-administration of MR and TCV Arm E: Co-administration of MR and OCV Arm F: Co-administration of TCV and OCV

1. Visit 1: Day 0

   * After describing the study procedure to the parents/guardian, the study staff will confirm that the child is eligible to participate in the study. If the child is eligible, written informed consent will be obtained from the parents/guardian for the participation of their child in the study. If the parents/guardian provide consent, a participant identification number (PID) will be assigned for the child.
   * Relevant demographic and clinical information of the participants will be captured in the eCRF.
   * Collect a blood sample (2-3 ml) from the child through venipuncture.
   * Allocate the study participant to the study group through a randomized process as described above.
   * Administration of the 1st dose of the study vaccines as per designated study arm (Table 1). Regarding co-administration of two vaccines, the participants will be observed for 30 minutes to monitor for any immediate adverse reactions or any anaphylaxis reaction after each vaccination.
   * The participants and their parents/guardians will be informed about the next schedule visit. They will also be asked to contact immediately if any adverse events occur within 7 days of vaccination.
2. Visit 2: Day 28 (+7)

   * Participant's clinical information including presence of diarrhea, fever and receipt of other vaccines will be captured in the eCRF.
   * Collect a blood sample (2-3 ml) from the child through venipuncture
   * Second dose of OCV vaccine will be given for the children of A (OCV only), E (MR + OCV) and F (TCV + OCV)
   * Observe the child for 30 minutes to monitor for any immediate adverse reactions or any anaphylaxis reaction to the vaccine.
   * The participants and their parents/guardians will be informed about the next schedule visit. They will also be asked to contact immediately if any adverse events occur within 7 days of vaccination.
3. Visit 3: Day 56 (+7)

   * Participant's clinical information including presence of diarrhea, fever and receipt of other vaccines will be captured in the eCRF.
   * Collect a blood sample (2-3 ml) from the child through venepuncture for arms A (OCV only), E (MR + OCV) and F (TCV + OCV)
   * First dose of MR vaccine will be given for the children of arms A (OCV only), B (TCV only) and F (TCV + OCV)
   * Observe the child for 30 minutes to monitor for any immediate adverse reactions or any anaphylaxis reaction to the vaccine.
   * The participants and their parents/guardians will be informed about the next schedule visit. They will also be asked to contact immediately if any adverse events occur within 7 days of vaccination.
4. Visit 4: Day 84 (+7)

   * Participant's clinical information including presence of diarrhea, fever and receipt of other vaccines will be captured in the eCRF.
   * Collect a blood sample (2-3 ml) from the child through venipuncture for arms A (OCV only), B (TCV only) and F (TCV + OCV)
   * The participants and their parents/guardians will be informed about the next schedule visit.
5. Visit 5: Day 180 (+7)

   * Participant's clinical information including presence of diarrhea, fever and receipt of other vaccines will be captured in the eCRF.
   * Second dose of MR vaccine will be given for the children of arms C (MR only), D (MR + TCV) and E (MR + OCV)
   * Observe the child for 30 minutes to monitor for any immediate adverse reactions or any anaphylaxis reaction to the vaccine.
   * The participants and their parents/guardians will be informed about the next schedule visit. They will also be asked to contact immediately if any adverse events occur within 7 days of vaccination.
6. Visit 6: Day 208 (+7):

   * Participant's clinical information including presence of diarrhea, fever and receipt of other vaccines will be captured in the eCRF.
   * Collect a blood sample (2-3 ml) from the child through venipuncture arms C (MR only), D (MR + TCV) and E (MR + OCV)
   * The participants and their parents/guardians will be informed about the next schedule visit.
7. Visit 7: Day 236 (+7)

   * Participant's clinical information including presence of diarrhea, fever and receipt of other vaccines will be captured in the eCRF.
   * Second dose of MR vaccine will be given for the children of arms A (OCV only), B (TCV only) and F (OCV + TCV)
   * Observe the child for 30 minutes to monitor for any immediate adverse reactions or any anaphylaxis reaction to the vaccine.
   * The participants and their parents/guardians will be informed about the next schedule visit. They will also be asked to contact immediately if any adverse events occur within 7 days of vaccination.
8. Visit 8: Day 264 (+7)

   * Participant's clinical information including presence of diarrhea, fever and receipt of other vaccines will be captured in the eCRF.
   * Collect a blood sample (2-3 ml) from the child through venipuncture arms A (OCV only), B (TCV only) and F (OCV + TCV)

Laboratory assay:

Vibriocidal assay Serum vibriocidal antibodies to V. cholerae O1 (El Tor Inaba; strain T19479; El Tor Ogawa; strain X25049) will be evaluated by a microtitre assay. The vibriocidal titre will be defined as the highest dilution causing 50% inhibition of bacterial growth. Two-fold serial dilutions of different day points specimens will be tested side-by-side in duplicates on each plate. Titres will be adjusted in relation to a reference serum specimen included in each test to compensate for variations between analyses on different occasions. The vibriocidal antibody titre ascribed to each sample will be the mean of the duplicated determinations, which will not be allowed to vary more than one two-fold dilution for either the reference or the test sera. The tests will be repeated if larger variations are observed. A four-fold or greater increase in titre between pre- and post-immunization specimens will be taken to represent seroconversion. To control for variations, test plates will contain pooled convalescent serum sample from patients with cholera as a positive control (pooled O1 Ogawa and O1 Inaba from our collection of specimens from cholera patients). Both positive and negative controls will be used, and all samples will be tested in triplicate.

The Vibriocidal assay will be carried out for the participants of arms A (OCV only), E (MR+OCV), and F (TCV+OCV) on days 0, 28, and 56.

Anti-Vi-IgG antibody measurement Blood samples will be transported to the laboratory to processed and stored by trained study staff, in accordance with standard operating procedures (SOP). The plasma/serum will be stored and used to measure the induced immune response in the vaccinee. The primary laboratory technique performed will be anti-Vi antibody ELISA performed on the extracted plasma sample, using a commercially available assay (VaccZyme, The Binding Site). This assay will be performed according to the manufacturer's instructions.

The assay will be carried out for the participants of arms of B (TCV only), D (MR+TCV), and F (TCV+OCV) on days 0, and 28

Measles and Rubella IgG antibody titres Measles antibody (IgG) will be measured using commercially available Enzyme-linked Immunosorbent Assay (ELISA) kits (Hycor Biomedical GmbH, Kassel, Germany or any other available kits). Anti-rubella IgG will also be detected using ELISA kit from Diasorin s.r.l., Italy or any other available kits. A standard curve run for each assay and quantitative values will be determined extrapolating the curve. Negative and positive controls (respective human sera will be supplied with the kit) will be run for each assay as quality control of the assay. The cut-off level of IgG antibody, protective and non-protective level for MR was determined according to the manufacturer's guidelines.

The assay will be carried out for the participants of arms A (OCV only), B (TCV only), C (MR only), D (MR+TCV), E (MR+OCV), and F (TCV+OCV) (days 0, 84, and 264 for the arms of A, B, and F; and days 0, 28, and 208 for the arms of C, D, and E).

Definition of seroconversion Seroconversion for typhoid (TCV): ≥4-fold rise of anti-Vi IgG antibody titres from day 0 to 28 days after receipt of TCV.

Seroconversion for cholera : ≥4-fold rise of vibriocidal antibody titres from day 0 to 28 days after receipt of first and second doses of OCV.

Seroconversion for measles and rubella vaccine:

≥4-fold rise of IgG antibody titer from day 0 to 28 days after receipt of first and second doses of measles and rubella vaccine. Specimens lacking detectable antibody before vaccination that will have antibody after vaccination will be considered as seroconversion.

Safety reporting:

Safety Monitoring After the 30 minutes observation period for anaphylactic reactions, the study physicians will record the presence of any potential reaction to the vaccine on the corresponding CRF.

Recording, Monitoring and Reporting of Adverse Events During each study clinic visit, study staff will question the parents about possible adverse events (AE) experienced by the participant since the previous study visit. This information will be recorded on the corresponding CRF. Reported AE will be recorded in the AE form. The AE form will include a description of the event, time of onset, assessment of severity, relationship to study product, and time of resolution/stabilization of the event. The adverse event reporting period will be for 7 days after each dose of any of the vaccines.

A 4-5 member data safety and monitoring board (DSMB) will be constructed for this project by the ERC of the icddr,b. This will be comprised of members of the ERC, staff members of icddr,b, and individuals from other institutions in Bangladesh. The DSMB members will not be involved in the study in any way.

The main responsibility of DSMB is to review the collected AEs under blinded or unblinded and evaluate the safety, provide recommendations on trial execution, and adjustments to the sponsor based on the analysis results.

Interpretation of vaccine-relationship to AE will be based on the type of event, the relationship of the event to the time of vaccine administration, the known biology of the vaccine, and the investigators' medical judgment.

All SAEs, occurring within the first 30 days of post vaccine administration, will be reported to the DSMB within 24 hours of notification. A more detailed report form will be completed including medical follow-up, and sent to the DSMB within the shortest period.

After 30 days of post vaccination, all SAEs will be recorded in the CRFs over the study period. The participant will be followed by a medically qualified investigator either until resolution, or until the event is considered as stable.

Sample size calculation and outcome:

The investigators propose to conduct an open-label, randomized controlled, non-inferiority study of co-administration of MR, OCV and TCV vaccination among children 12 to 59 months of age in Dhaka, Bangladesh. Children who did not receive any of the aforementioned vaccines will be included in the study. The number of children needed in each study arm will vary, with the sample size for each co-administration arm determined by the more conservative estimate (i.e. the larger of the two sample sizes required for the component vaccines). For MR, assuming that the percentage of children who will seroconvert for MR is approximately 75% for measles and 95% for rubella, a non-inferiority margin of 10%, and 20% attrition rate, 250 children per group will be required for 80% power and 97.5% one-sided confidence level. For OCV, assuming that the percentage of children who will seroconvert for OCV is approximately 70%, a non-inferiority margin of 10% and 20% attrition rate, 413 children per group will be required for 80% power and 97.5% one-sided confidence level. For TCV, assuming that the percentage of children who will seroconvert for TCV is approximately 80%, a non-inferiority margin of 10% and 20% attrition rate, 314 children per group will be required for 80% power and 97.5% one-sided confidence level. A total of 2117 children will be assigned in different arms based on the sample size calculation.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed written consent from participants parent/legal guardian
2. Participants aged 12 months to 59 months
3. Family does not have any plan to move from the study area during study period
4. No history of receipt of MR (Measles and Rubella) or TCV or OCV

Exclusion Criteria:

1. Child live outside of the study area
2. Participant with confirmed or suspected immunosuppressive or immunodeficiency disorder; or participant on any immunosuppressive or immunostimulant therapy
3. Known case of thrombocytopenia or any coagulation disorder, or participant on anticoagulation therapy
4. History of hypersensitivity reaction to any component of the study vaccines
5. Participant with febrile illness (temperature >37.9oC) at the time of enrollment
6. Participant with acute diarrhea and/or vomiting at the time of enrollment
7. Participant with acute infection or illness at the time of enrollment
8. Participant is severely malnourished

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2117 (Estimated)
Dates: Start 2023-10-14 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Vibriocidal antibody response for OCV | Two months
  * Vibriocidal antibody response for OCV when administered individually versus when co-administered with TCV on days 28 and 56
  * Vibriocidal antibody response for OCV when administered individually versus when co-administered with MR on days 28 and 56
Seroconversion for TCV | One Year
  * Seroconversion (≥4 fold rise of anti-Vi-IgG antibody titres compared to pre-vaccination) for TCV when administered individually versus when co-administered with OCV on day 28
  * Seroconversion (≥4 fold rise of anti-Vi-IgG antibody titres compared to pre-vaccination) for TCV when administered individually versus when co-administered with MR on day 28
Seroconversion for MR vaccine | One year
  * Seroconversion (≥4 fold rise of measles IgG antibody titres compared to pre-vaccination) for MR when administered individually versus when co-administered with OCV on days 28 and 208
  * Seroconversion (≥4 fold rise of measles IgG antibody titres compared to pre-vaccination) for MR when administered individually versus when co-administered with TCV on days 28 and 208
  * Seroconversion (≥4 fold rise of measles IgG antibody titres compared to pre-vaccination) for MR when administered individually versus when administered after OCV on days 84 and 264
Safety: number of adverse events and serious adverse events | One year
  Number of adverse events and serious adverse events when OCV, TCV and MR vaccines are co-administered versus given alone.

CONTACTS AND LOCATIONS:
Overall Officials: Md Taufiqul Islam, MBBS, MPH, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harapan H, Shields N, Kachoria AG, Shotwell A, Wagner AL. Religion and Measles Vaccination in Indonesia, 1991-2017. Am J Prev Med. 2021 Jan;60(1 Suppl 1):S44-S52. doi: 10.1016/j.amepre.2020.07.029. Epub 2020 Nov 12. PMID 33189503
- [Background] Dabbagh A, Patel MK, Dumolard L, Gacic-Dobo M, Mulders MN, Okwo-Bele JM, Kretsinger K, Papania MJ, Rota PA, Goodson JL. Progress Toward Regional Measles Elimination - Worldwide, 2000-2016. MMWR Morb Mortal Wkly Rep. 2017 Oct 27;66(42):1148-1153. doi: 10.15585/mmwr.mm6642a6. PMID 29073125
- [Background] Vynnycky E, Adams EJ, Cutts FT, Reef SE, Navar AM, Simons E, Yoshida LM, Brown DW, Jackson C, Strebel PM, Dabbagh AJ. Using Seroprevalence and Immunisation Coverage Data to Estimate the Global Burden of Congenital Rubella Syndrome, 1996-2010: A Systematic Review. PLoS One. 2016 Mar 10;11(3):e0149160. doi: 10.1371/journal.pone.0149160. eCollection 2016. PMID 26962867
- [Background] Ali M, Nelson AR, Lopez AL, Sack DA. Updated global burden of cholera in endemic countries. PLoS Negl Trop Dis. 2015 Jun 4;9(6):e0003832. doi: 10.1371/journal.pntd.0003832. eCollection 2015. PMID 26043000
- [Background] Islam MT, Clemens JD, Qadri F. Cholera Control and Prevention in Bangladesh: An Evaluation of the Situation and Solutions. J Infect Dis. 2018 Oct 15;218(suppl_3):S171-S172. doi: 10.1093/infdis/jiy470. No abstract available. PMID 30169839
- [Background] Mogasale V, Maskery B, Ochiai RL, Lee JS, Mogasale VV, Ramani E, Kim YE, Park JK, Wierzba TF. Burden of typhoid fever in low-income and middle-income countries: a systematic, literature-based update with risk-factor adjustment. Lancet Glob Health. 2014 Oct;2(10):e570-80. doi: 10.1016/S2214-109X(14)70301-8. PMID 25304633
- [Background] Chowdhury F, Bhuiyan TR, Akter A, Bhuiyan MS, Khan AI, Hossain M, Tauheed I, Ahmed T, Islam S, Rafique TA, Siddique SA, Harun NB, Islam K, Clemens JD, Qadri F. Immunogenicity of a killed bivalent whole cell oral cholera vaccine in forcibly displaced Myanmar nationals in Cox's Bazar, Bangladesh. PLoS Negl Trop Dis. 2020 Mar 16;14(3):e0007989. doi: 10.1371/journal.pntd.0007989. eCollection 2020 Mar. PMID 32176695
- [Background] Chowdhury F, Bhuiyan TR, Akter A, Bhuiyan MS, Khan AI, Tauheed I, Ahmed T, Ferdous J, Dash P, Basher SR, Hakim A, Lynch J, Kim JH, Excler JL, Kim DR, Clemens JD, Qadri F. Augmented immune responses to a booster dose of oral cholera vaccine in Bangladeshi children less than 5 years of age: Revaccination after an interval of over three years of primary vaccination with a single dose of vaccine. Vaccine. 2020 Feb 11;38(7):1753-1761. doi: 10.1016/j.vaccine.2019.12.034. Epub 2019 Dec 24. PMID 31879124
- [Background] Qadri F, Khanam F, Liu X, Theiss-Nyland K, Biswas PK, Bhuiyan AI, Ahmmed F, Colin-Jones R, Smith N, Tonks S, Voysey M, Mujadidi YF, Mazur O, Rajib NH, Hossen MI, Ahmed SU, Khan A, Rahman N, Babu G, Greenland M, Kelly S, Ireen M, Islam K, O'Reilly P, Scherrer KS, Pitzer VE, Neuzil KM, Zaman K, Pollard AJ, Clemens JD. Protection by vaccination of children against typhoid fever with a Vi-tetanus toxoid conjugate vaccine in urban Bangladesh: a cluster-randomised trial. Lancet. 2021 Aug 21;398(10301):675-684. doi: 10.1016/S0140-6736(21)01124-7. Epub 2021 Aug 9. PMID 34384540
- [Background] Tischer A, Andrews N, Kafatos G, Nardone A, Berbers G, Davidkin I, Aboudy Y, Backhouse J, Barbara C, Bartha K, Bruckova B, Duks A, Griskevicius A, Hesketh L, Johansen K, Jones L, Kuersteiner O, Lupulescu E, Mihneva Z, Mrazova M, De Ory F, Prosenc K, Schneider F, Tsakris A, Smelhausova M, Vranckx R, Zarvou M, Miller E. Standardization of measles, mumps and rubella assays to enable comparisons of seroprevalence data across 21 European countries and Australia. Epidemiol Infect. 2007 Jul;135(5):787-97. doi: 10.1017/S0950268807008266. Epub 2007 Mar 30. PMID 17394675
- [Background] Sirima SB, Ouedraogo A, Barry N, Siribie M, Tiono A, Nebie I, Konate A, Berges GD, Diarra A, Ouedraogo M, Bougouma EC, Soulama I, Hema A, Datta S, Liang Y, Rotrosen ET, Tracy JK, Jamka LP, Oshinsky JJ, Pasetti MF, Neuzil KM, Laurens MB. Safety and immunogenicity of Vi-typhoid conjugate vaccine co-administration with routine 9-month vaccination in Burkina Faso: A randomized controlled phase 2 trial. Int J Infect Dis. 2021 Jul;108:465-472. doi: 10.1016/j.ijid.2021.05.061. Epub 2021 Jun 1. PMID 34082090
- [Background] Chowdhury F, Ali Syed K, Akter A, Rahman Bhuiyan T, Tauheed I, Khaton F, Biswas R, Ferdous J, Al Banna H, Ross AG, Mc Millan N, Sharma T, Kanchan V, Pal Singh A, Gill D, Lebens M, Nordqvist S, Holmgren J, Clemens JD, Qadri F. A phase I/II study to evaluate safety, tolerability and immunogenicity of Hillchol(R), an inactivated single Hikojima strain based oral cholera vaccine, in a sequentially age descending population in Bangladesh. Vaccine. 2021 Jul 22;39(32):4450-4457. doi: 10.1016/j.vaccine.2021.06.069. Epub 2021 Jul 1. PMID 34218960
- [Background] Redd SC, King GE, Heath JL, Forghani B, Bellini WJ, Markowitz LE. Comparison of vaccination with measles-mumps-rubella vaccine at 9, 12, and 15 months of age. J Infect Dis. 2004 May 1;189 Suppl 1:S116-22. doi: 10.1086/378691. PMID 15106100
- [Background] Saha A, Chowdhury MI, Khanam F, Bhuiyan MS, Chowdhury F, Khan AI, Khan IA, Clemens J, Ali M, Cravioto A, Qadri F. Safety and immunogenicity study of a killed bivalent (O1 and O139) whole-cell oral cholera vaccine Shanchol, in Bangladeshi adults and children as young as 1 year of age. Vaccine. 2011 Oct 26;29(46):8285-92. doi: 10.1016/j.vaccine.2011.08.108. Epub 2011 Sep 9. PMID 21907255